CLINICAL TRIAL: NCT06513728
Title: Methadone Patient Access to Collaborative Treatment
Brief Title: Pilot Study of Methadone Patient Access to Collaborative Treatment: a HEAL Initiative
Acronym: MPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 456482
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: Opioid Substitution Treatment Clinics; Patients; Staff
Keywords: Implementation Science; Methadone treatment; Opioid Use Disorder; Opioid Use Disorder Treatment; Workforce Development; Vicarious trauma; Posttraumatic stress; Treatment retention
MeSH Terms: conditions — Opioid-Related Disorders; Compassion Fatigue

STUDY DESIGN:
Intervention Model Description: This is a pilot implementation and preliminary effectiveness study of MPACT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MPACT Intervention (Experimental): Single arm study. All sites will receive the intervention.
  Interventions: Other: MPACT Intervention

INTERVENTIONS:
Other: MPACT Intervention — MPACT has 4 components: accredited training about patient centered, trauma informed methadone treatment, staff education about trauma symptoms with navigation to self screening and treatment or stress management, clinic self assessment tools for trauma informed, patient centered care, and reflective supervision for counselors, case managers and peer staff.

SUMMARY:
Examine the preliminary effect of the MPACT intervention on methadone treatment retention, in treatment overdose and patient trauma symptoms. The study will also explore the relationship between staff trauma symptoms and MPACT implementation.

DETAILED DESCRIPTION:
Specific AIMS:

AIM 1: Develop MPACT through multilevel, iterative planning with OTP staff and people with recent MMT experience.

AIM 2: Conduct a 4-month MPACT pilot test in two AZ OTPs: Mesa (urban) with 50 patients and 22 staff, and Sierra Vista (rural-serving) with 50 patients and 8 staff to:

1. Determine MPACT implementation feasibility, acceptability, and preliminary effect on MMT practice change and culture.
2. Determine MPACT preliminary effect on MMT retention, in-MMT overdose, and patient PTSS.
3. Characterize staff trauma history, PTSS and vicarious trauma, and explore their relationship with MPACT acceptability and implementation fidelity.

AIM 3: Characterize MPACT acceptability, likely adoption, and recruitment feasibility among directors, case managers and counselors from a national random sample of 500 OTPs.

ELIGIBILITY:
Inclusion Criteria:

* Staff of enrolled opioid treatment programs (methadone clinics) who are involved with methadone treatment
* Patients receiving methadone at these locations

Exclusion Criteria:

* Patients not receiving methadone at these locations
* Staff not involved in methadone treatment at these locations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
methadone treatment retention | 4 months (pilot study period)
  Retention in methadone treatment (measured by 3 different indicators)
In treatment overdose | 4 months (pilot study period)
  Reported overdoses during methadone treatment (measured by study constructed algorithm)

SECONDARY OUTCOMES:
Trauma symptoms among patients and staff | pilot period of 4 months
  Post traumatic stress symptoms (measured by 8-item Post Traumatic Stress Disorder Checklist or, PCL-5). Scores are 0-80. Higher scores mean greater PTSD symptom severity.
Vicarious Trauma symptoms among staff | pilot period of 4 months
  Vicarious trauma symptoms (measured by the Vicarious Trauma Scale (VTS). Scores are 0-190. Higher scores indicate more vicarious (work related) traumatization.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Meyerson, PhD, Principal Investigator — Professor
Locations (1):
- University of Arizona College of Medicine, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
A Data Sharing and Management Plan was submitted to NIDA for this study. please see that submission.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 1 year after the study completion
Access Criteria: See Data sharing and management plan

REFERENCES:
- [Derived] Meyerson BE, Davis A, Crosby RA, Linde-Krieger LB, Brady BR, Carter GA, Mahoney AN, Frank D, Rothers J, Coffee Z, Deuble E, Ebert J, Jablonsky MF, Juarez M, Lee B, Lorenz HM, Pava MD, Tinsely K, Yousaf S. Methadone Patient Access to Collaborative Treatment: Protocol for a Pilot and a Randomized Controlled Trial to Establish Feasibility of Adoption and Impact on Methadone Treatment Delivery and Patient Outcomes. JMIR Res Protoc. 2025 Apr 15;14:e69829. doi: 10.2196/69829. PMID 40105313